CLINICAL TRIAL: NCT03991832
Title: A Phase II Study of Olaparib and Durvalumab (MEDI 4736) in Patients With IDH-Mutated Solid Tumors
Brief Title: Study of Olaparib and Durvalumab in IDH-Mutated Solid Tumors
Acronym: SOLID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-5526; SOLID (Other: Princess Margaret Cancer Centre)
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Glioma; Cholangiocarcinoma; Solid Tumor; IDH Mutation
MeSH Terms: conditions — Glioma; Cholangiocarcinoma | interventions — olaparib; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: IDH mutated glioma (Experimental): Olaparib, by mouth (orally), twice a day, every day. Durvalumab, by vein (intravenously), on Day 1 of every 28 day cycle.
  Interventions: Drug: Olaparib; Drug: Durvalumab
- Cohort B: IDH mutated cholangiocarcinoma (Experimental): Olaparib, by mouth (orally), twice a day, every day. Durvalumab, by vein (intravenously), on Day 1 of every 28 day cycle.
  Interventions: Drug: Olaparib; Drug: Durvalumab

INTERVENTIONS:
Drug: Olaparib — Olaparib is a drug that blocks a protein called poly (ADP-ribose) polymerase (PARP). PARP is important in the growth and spread of cancer cells. Because of this, blocking PARP from working is expected to stop the growth of or shrink cancer cells.
  Other Names: Lynparza
Drug: Durvalumab — Durvalumab is a drug that works by stopping a protein called Programmed Cell Death Ligand 1 (PD-L1) from working. PD-L1 is a protein that is thought to prevent the immune system (the body's defense against diseases) from killing cancer cells. Stopping PD-L1 from working is expected to allow the immune system to once again prevent or slow down cancer growth.
  Other Names: Imfinzi

SUMMARY:
This is a phase 2 study of the combination of drugs olaparib and durvalumab for the treatment of isocitrate dehydrogenase or (IDH) mutated solid tumors. The purpose of this study is to assess the efficacy of the drug combination via overall response rate and overall disease control rate.

It is believed that giving olaparib and durvalumab together would be more useful when given to patients with IDH-mutated solid tumors than giving each drug alone.

DETAILED DESCRIPTION:
Patients with documented IDH mutations will be screened for eligibility within 4 weeks of the start of study treatment including medical history, physical exam, height, weight, vital signs, performance status, routine blood lab tests, pregnancy test, ECG, and tumor measurements for safety, and research blood and archival tumor tissue collection for biomarker research. In the event participants require surgery or biopsy during their participation in the study, samples of the tumor tissue removed will be collected for biomarker research.

Eligible participants will be assigned to a cohort depending on their type of cancer:

* Cohort A: IDH-mutated glioma (a type of brain/spinal cord cancer)
* Cohort B: IDH-mutated cholangiocarcinoma (a type of bile duct cancer)

While on the study drugs, participants will have many of the screening tests and procedures repeated for safety and for biomarker research.

If participants are permanently taken of the study drugs for any reason, they will be asked to return to the clinic about 4 weeks after the last dose of study drugs to have tests and procedures done during the study repeated for safety and research purposes.

After the End of Study Drug visit, participants will continue to be followed-up by telephone or by clinic visit every 8-12 weeks until they no longer wish to be followed or start a new anti-cancer treatment, or until 1 year after last dose of study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Must be ≥ 18 years.
* Body weight > 30 kg.
* For Cohort A: Patients must have histologically or cytologically confirmed diffuse astrocytic and oligodendroglial tumors by World Health Organization 2016 classification which are IDH mutant. They must have not received more than 2 regimens of systemic therapy after initial relapse.
* For Cohort B: Patients must have histologically or cytologically confirmed adenocarcinoma of the biliary tract which are IDH mutant. They must have not received more than 2 regimens of systemic therapy for advanced disease.
* Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must have a life expectancy ≥ 16 weeks.
* All participants must agree to use methods to prevent pregnancy as agreed upon between the participant and the study doctor from the signing of the informed consent form and continue throughout the period of taking study treatments and for 3 months after the last doses of study drugs.
* Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Patients in Cohorts A and B must have measurable disease
* Patients with glioma or central nervous system (CNS) metastases must be asymptomatic and at least 28 days after the most recent CNS treatment and is clinically stable, and at least 14 days on stable doses of corticosteroids and/or anti-seizure medications.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study.
* Concurrent enrolment in another clinical study, unless it is an observational (non-intervention) clinical study or the follow-up period of an interventional study.
* Receipt of any conventional or investigational anticancer therapy within 4 weeks prior to the planned first dose of olaparib and durvalumab.
* Any previous treatment with PARP inhibitor or PD-1/PD-L1 inhibitors including olaparib and durvalumab.
* Other malignancy within the last 5 years with exceptions.
* Resting ECG with QTc > 470 msec or family history of long QT syndrome.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 4 weeks prior to planned start of study treatment.
* Concomitant use of known strong or moderate CYP3A inducers. The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents. This criterion does not apply to patients in Cohort A.
* Persistent toxicities caused by previous cancer therapy, excluding alopecia and laboratory values listed per the inclusion criteria.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients with symptomatic uncontrolled brain metastases.
* Major surgery within 2 weeks of starting study treatment. Patients must have recovered from any effects of any major surgery to be considered eligible.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of olaparib.
* Female patients who are pregnant, lactating, or intend to become pregnant during their participation in this study.
* Immunocompromised patients.
* Patients with a known hypersensitivity to olaparib or durvalumab or any of the excipients of the products.
* Patients with known active hepatitis (i.e. Hepatitis B or C).
* Patients requiring whole blood transfusions in the last 120 days prior to entry to the study.
* Current or prior use of immunosuppressive medications within 14 days before the 1st dose with exceptions.
* Active or prior documented autoimmune or inflammatory disorders within the last 2 years.
* History of allogenic organ transplantation.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational products or interpretation of patient safety or study results.
* Prior enrolment in this study.
* Receipt of liver attenuated vaccines within 30 days prior to the 1st dose of investigational products, during the study and 30 days after the last dose of study treatments.
* Known active infection including tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 3 years
  overall + partial response
Overall disease control rate | 3 years
  for both cohorts

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  For duration of study
Overall survival | 3 years
  for duration of study
Number of incidences of adverse events | 3 years
  for duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Eric Chen, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No